CLINICAL TRIAL: NCT02047994
Title: Multicentric Randomized Study of H. Pylori Eradication and Pepsinogen Testing for Prevention of Gastric Cancer Mortality
Acronym: GISTAR
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: International Agency for Research on Cancer (Other)
Collaborators: University of Latvia (Other); Technion, Israel Institute of Technology (Other); Karolinska Institutet (Other); Academic Histology Laboratory (Latvia) (Other); Vanderbilt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12-36
Record Dates: First submitted 2014-01-27; First posted 2014-01-29 (Estimated); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Helicobacter Pylori Infections; Atrophic Gastritis; Gastric Cancer
Keywords: Gastric cancer; Gastric cancer mortality; Helicobacter pylori treatment; Pepsinogen testing; Endoscopy; Volatile marker
MeSH Terms: conditions — Gastritis, Atrophic; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1:Triple therapy (Experimental): Among those assigned to Group 1, participants who are Helicobacter pylori positive will receive Triple therapy and/or upper endoscopy. Participants with serological evidence of atrophic gastritis will undergo upper endoscopy and further endoscopic follow-up. H. pylori positive individuals will be offered Helicobacter pylori eradication as appropriate, independently of the pepsinogen results. From subjects in this group, breath samples will also be collected for volatile markers study. In addition, fecal occult blood test (FOBT) will be offered to this group as a benefit to participate in the study.
  Interventions: Drug: Triple therapy
- Group 2:No intervention (No Intervention): Those who assigned to Group 2 will receive no intervention and will be offered FOBT as a benefit of study participation. Any participants who show positive FOBT will be referred to colonoscopy. This will be the benefit to this group together with initial medical evaluation at the time of inclusion. During the follow-up period this group will be offered to consult a specialist when required due to clinical symptoms.

INTERVENTIONS:
Drug: Triple therapy — Participants who are positive with Helicobacter pylori in Group1 will receive triple therapy.
  * Esomeprazole 40 mg bid for 10 days
  * Clarithromycin 500 mg bid for 10 days
  * Amoxicillin 1000 mg bid for 10 days
  Arms: Group 1:Triple therapy

SUMMARY:
Currently no ideal preventive modalities are available for reducing gastric-cancer caused mortality in organized population-based application. The primary objective of the study is to determine if H.pylori screening followed by eradication of positive subjects and endoscopic follow-up of those with serological evidence of atrophic gastritis reduces mortality from gastric cancer in middle-aged people in high-risk areas. The GISTAR study is a multicenter randomized study of H.pylori eradication and pepsinogen testing for prevention of gastric cancer mortality. Altogether 30.000 individuals aged 40-64 years will be enrolled, providing 90% study power to detect at least 35% reduction in gastric cancer mortality at 15 years of follow-up. Participants will be randomly allocated to one of two groups. In the active investigation/management group those positive for H.pylori will be offered eradication therapy and individuals with decreased pepsinogen I/II ratio will be invited for endoscopy. The control group will receive standard health care. The primary endpoint for this trial will be the mortality difference from gastric cancer between the two groups at 15 years or when enough cases accumulate to demonstrate a statistical difference. The study is expected to provide valuable information on the utility for reduction in gastric cancer mortality of: 1) H.pylori eradication in adults on a population-basis, including subjects who may already have pre-malignant lesions; and 2) pepsinogen testing in screening settings. A pilot study of 3,455 individuals prior to the main trial was conducted from October 2013 to December 2016.

DETAILED DESCRIPTION:
Gastric cancer is an important global public health issue in Eastern European regions, where the burden of the disease is substantial. There is sufficient epidemiological and experimental evidence that supports a causal link between H. pylori and gastric cancer. However, there is still limited evidence from clinical trials to prove whether H. pylori eradication with antimicrobial therapy is the approach of choice in entire infected populations or only in selected groups to reduce the risk of gastric cancer and whether eradication at advanced stages of atrophy is effective among these patients. The current European and global guidelines are proposing screening with pepsinogen tests as the best available tool to identify the individuals at increased risk for cancer development, yet there is insufficient evidence available on how effective these tests are in organized cancer screening settings.

We therefore propose to conduct a multi-center randomized trial in Latvia, Belarus and Russia, areas with high burden of the disease, with the main objective of evaluating if H. pylori screening followed by eradication in participants with positive result and endoscopy of those with serological evidence of atrophic gastritis can reduce gastric cancer mortality. The proposed trial will also investigate retrospectively if groups with chronic atrophic gastritis can select subjects who require treatment to achieve comparable gastric cancer reduction. Ultimately, this study will have the potential to find effective prevention strategies through identifying appropriate target groups that could get most benefits from the treatment.

The aim of this study is to search for new intervention strategies to decrease mortality from gastric cancer in high-risk areas.

The primary objective of the study is to determine if H. pylori screening followed by eradication of positive subjects and endoscopic follow-up of those with serological evidence of atrophic gastritis reduces mortality from gastric cancer in a high risk population among 40-64 years old subjects.

The secondary objectives are:

1. To determine retrospectively if biomarkers of chronic atrophic gastritis or others can select the group of subjects who require treatment to achieve gastric cancer reduction comparable to the primary objective.
2. To evaluate the rationale for volatile marker testing in exhaled breath for early identification of lesions in the stomach as well as other conditions related to increased risk.
3. To evaluate the role of diet, lifestyle factors and environmental factors in the development of gastric lesions.
4. To evaluate the impact of H. pylori eradication on selected medical conditions potentially associated with the infection (e.g. obesity, inflammatory bowel disease, dementia, circulatory diseases and esophageal diseases)

Methods: Approximately 30,000 men and women will be recruited into a randomized study. Eligible subjects between 40-64 years of age at entry who are residents in high gastric cancer incidence areas will be invited to participate in the trial by visiting one of the study clinics set up specifically for this trial.

For eligible participants who agree to participate and sign informed consent, a risk factor questionnaire will be administered and a complete medical evaluation will be performed at baseline.

Participants will be randomly assigned to either Group 1 (50%) or Group 2 (50%). Among those assigned to Group 1, H. pylori screening by detecting immunoglobulin G (IgG) group antibodies in plasma/serum and pepsinogen test will be performed. According to the results of the tests, participants will be assigned to H. pylori eradication treatment or upper endoscopy. Participants with serological evidence of atrophic gastritis (low pepsinogen I/II ratio) will undergo upper endoscopy with appropriate biopsy sampling as well as further follow-up with endoscopy according to MAPS (Management of precancerous conditions and lesions in the stomach) guidelines. H. pylori positive individuals will be offered standard eradication treatment as appropriate. From subjects in this group, breath samples will also be collected for volatile markers study by research nurses or junior physicians.

Participants assigned to Group 2 (50%) will constitute the control group, after having had a medical evaluation at the time of recruitment. During the follow-up period this group will be offered to consult a specialist when required due to clinical symptoms.

Both Group 1 and Group 2 will be offered fecal occult blood test (FOBT) as a benefit of study participation. Any participants who show a positive FOBT result will be referred to colonoscopy.

All the trial participants including Group 2 will be followed up at least for 15 years to collect systematic information on medical conditions, in particular gastric cancer and cause of death. A follow-up telephone call /alternative communication will be made every 5 years for outcome assessment.

The general study is preceded by a pilot-study that was conducted from October 2013 to December 2016 to test the assumptions as well as the tools and functionality of the study infrastructure. According to the results of the pilot study, required infrastructure and tools planned in the general study will be adapted accordingly.

Endpoints: The primary endpoint for our trial will be the mortality difference from gastric cancer between Group 1 and Group 2 at 15 years or when enough cases accumulate to demonstrate a statistical difference between the groups.

In addition to the mortality difference from gastric cancer between the two groups, other endpoints required to achieve the secondary objectives are listed below:

* The difference in gastric cancer incidence between Group 1 and Group 2
* The all-cause mortality difference between Group 1 and Group 2
* The difference in incidence and mortality of medical conditions between Group 1 and Group 2
* Sensitivity and specificity of pepsinogen tests to detect atrophy
* The proportion of gastric cancers arising in patients with non-atrophic vs. atrophic gastritis
* The proportion of cancers arising in patients with atrophy, but negative for H. pylori infection
* The difference in incidence of gastric cancer in the group with successful eradication when compared to those refusing/failing eradication within Group I
* The proportion of gastric cancer cases being identified during scheduled follow-up endoscopy out of the total number of cases in the follow-up group
* The differences in the test performance and disease prevalence between ethnic groups
* The performance (sensitivity, specificity, overall accuracy) of volatile marker testing approach to diagnose gastric cancer as well as premalignant lesions in the stomach

A pilot study with 3,455 participants was started in October 2013 and completed in December 2016 in Latvia.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 40-64 at the time of signing the consent form
* Willingness to get involved in the study irrespective in which of the study arms (after detailed information on the potential benefits and risks that this study may confer)
* The person has signed a consent form (including the acceptance of transporting the samples over the borders, as appropriate)
* To be in good health, as determined by a physical examination and history performed by a study physician at enrolment

Exclusion Criteria:

* Personal history of gastric cancer (prevalent gastric cancer cases will not be revealed at the time of inclusion, and therefore will be included)
* Gastric resections due to benign disease (ulcer suturing and vagotomy are accepted)
* H. pylori eradication therapy within 12 months prior to inclusion (irrespective of the treatment result)
* Presence of alarm symptoms for digestive or any other diseases (detailed in the questionnaire or during the physician evaluation)
* Pathological findings at physical investigation suggestive for a serious organic disease (physician evaluation)
* Serious co-morbid condition with life expectancy less than 5 years (physician evaluation)
* Factors otherwise limiting the participation according to the protocol conditions (problems of mobility, etc.)
* Serious psychological conditions/psychiatric disease limiting the possibilities to understand the requirements for diagnostic and/or medical interventions (physician evaluation)
* Low expectations on the compliance for the diagnostic work-up or treatment (physician evaluation)
* Expected loss for the follow-up (e.g. lack of communication possibilities and data entry in the registries, expected travel abroad, etc.) (physician evaluation)
* Signed consent form is not available

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30000 (Estimated)
Dates: Start 2013-03 (Actual); Primary Completion 2033-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Gastric cancer mortality | 15 years
  The primary objective of the study is to determine if H. pylori screening followed by eradication of positive subjects and endoscopic follow-up of those with serological evidence of atrophic gastritis reduces mortality from gastric cancer in a high risk population among 40-64 years old subjects.

SECONDARY OUTCOMES:
Gastric cancer incidence | 15 years
  The difference in gastric cancer incidence between Group 1 and Group 2 will be investigated
All-cause mortality | 15 years
  The all-cause mortality difference between Group 1 and Group 2 will also be investigated.
Incidence of- and mortality from other medical conditions | 15 years
  The impact of H. pylori eradication on selected medical conditions potentially associated with the infection (e.g. obesity, inflammatory bowel disease, dementia, circulatory diseases and esophageal diseases) will be explored.

CONTACTS AND LOCATIONS:
Overall Officials: Marcis Leja, MD, PhD, Principal Investigator — Professor, Institute of Clinical and Preventive Medicine, University of Latvia; Jin Young Park, PhD, Principal Investigator — Early Detection, Prevention and Infections Branch, International Agency for Research on Cancer
Locations (1):
- Institute of Clinical and Preventive Medicine, University of Latvia, Riga, Latvia

REFERENCES:
- [Derived] Leja M, Cine E, Polaka I, Daugule I, Murillo R, Parshutin S, Razuka-Ebela D, Rotberga L, Anarkulova L, Krike P, Santare D, Tzivian L, Herrero R, Park JY. Factors influencing participation in preventive interventions for gastric cancer: the results from the GISTAR study. Eur J Cancer Prev. 2022 Mar 1;31(2):128-136. doi: 10.1097/CEJ.0000000000000682. PMID 34519690
- [Derived] Leja M, Park JY, Murillo R, Liepniece-Karele I, Isajevs S, Kikuste I, Rudzite D, Krike P, Parshutin S, Polaka I, Kirsners A, Santare D, Folkmanis V, Daugule I, Plummer M, Herrero R. Multicentric randomised study of Helicobacter pylori eradication and pepsinogen testing for prevention of gastric cancer mortality: the GISTAR study. BMJ Open. 2017 Aug 11;7(8):e016999. doi: 10.1136/bmjopen-2017-016999. PMID 28801429
- See also: Study official website — https://www.gistar.eu/